CLINICAL TRIAL: NCT04249024
Title: Comparing Treatment of Peri-implantitis With Either 970 nm Laser or Conventional Mucosal Flap Surgery - a Prospective Randomized Controlled Trial
Brief Title: Peri-implantitis, Comparing Treatments 970 nm Laser and Mucosal Flap Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Annsofi Johannsen, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Peri-implantitis 970 nm laser
Record Dates: First submitted 2019-10-16; First posted 2020-01-30 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Peri-Implantitis
Keywords: Peri-implantitis; Laser treatment; Surgical treatment; Randomized controlled trial; Patient reported outcomes; Clinical outcomes; Microbiology; Immunology
MeSH Terms: conditions — Peri-Implantitis | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Masking for the assessors of microbial, immunological and radiographic analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser treatment (Experimental): Laser treatment with diode laser 970nm and settings 1.2W in intervals of max 20s, until satisfactory removal of diseased epithelium and granulation tissue.
  Interventions: Device: Laser treatment; Behavioral: Oral hygiene instructions
- Mucosal flap surgery (Active Comparator): Conventional mucosal flap surgery of affected dental implant.
  Interventions: Procedure: Mucosal flap surgery; Behavioral: Oral hygiene instructions

INTERVENTIONS:
Device: Laser treatment — The participants in the laser group are treated with a 970 nm diode laser and if calculus is present scaling and root planning (SRP). The peri-implant pocket will be radiated with the 970 nm laser, removing bacteria, diseased epithelium and granulation tissue. The laser will be used at a maximum of 20s intervals before water irrigation. Laser settings continuous wave mode and power between 1.0-1.3W. Total treatment time will vary with the depth of the pocket and size of the surrounding bone crater.
  Arms: Laser treatment
Procedure: Mucosal flap surgery — The participants will receive a conventional peri-implant mucosal flap surgery of affected implants, and return after 7-10 days for suture removal. The surgery is a well-established treatment of peri-implantitis.
  Arms: Mucosal flap surgery
Behavioral: Oral hygiene instructions — Oral hygiene instructions of how to clean around dental implants as per individual needs in terms of access to clean and fine motor skills.

SUMMARY:
A clinical trial comparing laser treatment and conventional mucosal flap surgery for treatment of peri-implantitis. The main aim of the study is to evaluate if treatment of peri-implantitis with 970 nm laser combined with scaling and root planning (SRP) is clinically comparable to conventional mucosal flap surgery in terms of pocket probing depth reduction.

DETAILED DESCRIPTION:
The present project aims to evaluate a novel method in treating peri-implantitis, with focus on decreasing the patient's suffering as well as disease progression. Peri-implantitis has a direct influence on both physical and psychological wellbeing and have been related to difficulty in chewing due to loss of implants, bad esthetic appearance as well as high costs. Therefore, it is of importance for the individual as well as for the society to thoroughly investigate any new treatment approaches.

The study is a prospective randomized clinical trial comparing laser treatment (test group) and conventional mucosal flap surgery (active control group). Assessment of clinical variables at baseline and after 6 months. Patient reported outcomes at baseline, directly after treatment and after 10 days.

Primary Objective:

To evaluate if treatment of peri-implantitis with 970 nm laser combined with scaling and root planning (SRP) is clinically comparable to conventional mucosal flap surgery in terms of pocket probing depth reduction.

Secondary Objectives:

* To evaluate other clinical and radiological variables connected to peri-implantitis and the inflammation surrounding the dental implant.
* To evaluate the patient experience of treatment of peri-implantitis.
* To evaluate the inflammatory and microbial response after laser treatment

ELIGIBILITY:
Inclusion Criteria:

* Signs of peri-implantitis around one or more dental implants. All criteria below need to be fulfilled for inclusion.

  * Presence of pocket probing depth (PPD) > 5 mm
  * Bleeding on probing/suppuration (BOP/Pus)
  * At least 2 mm loss of bone, visible on radiographs, after initial osseointegration.
* ≥ 18 years old.
* Patient able to understand Swedish.

Exclusion Criteria:

* Antibiotic treatment 6 months prior to baseline.
* Peri-implant treatment 6 months prior to baseline.
* Myocardial infarction 6 months prior to baseline.
* Previous radiation treatment in the affected jaw area.
* Previous i.v. bisphosphonate treatment.
* Moderate or severe impairment of cognitive function (e.g. dementia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Mean change in pocket probing depth (PPD) | 0-6 months
  Pocket probing depth (PPD) will be measured by a 1 mm graded pocket probe from the bottom of the peri-implant pocket to the marginal mucosa and will be registered on 4 surfaces surrounding the implant.

SECONDARY OUTCOMES:
Mean change in plaque index (PI) | 0-6 months
  Plaque index (PI) will be measured at 4 sites per implant and assessed as per cent of the total amount of measured implant surfaces.
Mean change in bleeding on probing (BOP) | 0-6 months
  BOP will be registered on 4 surfaces surrounding the implant after probing the peri-implant pocket with a pocket probe, up to 20 s after the provocation with the probe.
Mean change in presence of suppuration | 0-6 months
  Presence of suppuration will be registered on 4 surfaces surrounding the implant after probing the peri-implant pocket with a pocket probe, up to 20 s after the provocation with the probe.
Mean change in marginal bone level on radiographs | 0-6 months
  Measured on radiographs for a fixed point on the dental implant to the marginal bone level.
Mean change in inflammatory response in peri-implant crevicular fluid (PICF) | 0-6 months
  Analysis of inflammatory meditators in PICF will be performed by commercially available ELISAs or multiplex assays at base line and 6 months. The analytes of interest to be tested are mainly inflammatory cytokines, chemokines, growth factors, proteases, and molecules related to bone remodeling such as for IL-1β, MMP 8, TIMP-1, CSF-1, elastase activity, and RANK-L/OPG ratio.
Mean change in inflammatory response in saliva | 0-6 months
  Analysis of inflammatory meditators in stimulated saliva will be performed by commercially available ELISAs or multiplex assays at base line and 6 months. The analytes of interest to be tested are mainly inflammatory cytokines, chemokines, growth factors, proteases, and molecules related to bone remodeling such as for IL-1β, MMP 8, TIMP-1, CSF-1, elastase activity, and RANK-L/OPG ratio.
Composition of the subgingival microflora | 0-6 months
  The bacterial composition in the subgingival microflora will be analyzed by quantitative real-time Polymerase Chain Reaction (qPCR).
Mean change in patient reported outcome using the visual analogue scale (VAS) score | Baseline, directly after treatment, 10 days after and 6 months after treatment.
  Visual analogue scale (VAS) is used to record the patients pain, discomfort and satisfaction with the treatment. The patients mark their response on a 100 mm line, with low values being no feeling of pain, discomfort or satisfaction, and high values meaning maximum pain, discomfort or satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Annsofi Johannsen, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Danakliniken Specialist Dentistry, Danderyd, Stockholm County
  - Specialist Dentistry Clinic, Karolinska Institutet, Dept. of Dental Medicine, Huddinge, Stockholm County

IPD SHARING:
Plan to Share IPD: No